CLINICAL TRIAL: NCT03866811
Title: Targeting High Risk Teens in the Emergency Department: A User-Informed, Theory-Based Intervention Using Text Messaging to Reduce Teen Pregnancy
Brief Title: Reducing Teen Pregnancy in the Emergency Department
Acronym: ERICA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Lauren S. Chernick, Assistant Professor of Pediatrics in Emergency Medicine, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AAAR6781 (Part 2); 1K23HD096060-01 (NIH)
Record Dates: First submitted 2019-02-08; First posted 2019-03-07 (Actual); Results first posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-07

CONDITIONS: Reproductive Behavior; Sexual Behavior; Adolescent Behavior; Contraception
Keywords: emergency medicine; reproductive health; sexual health; adolescent health; emergency department; text messaging; mobile health; digital health
MeSH Terms: conditions — Reproductive Behavior; Sexual Behavior; Adolescent Behavior; Emergencies

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial with two arms
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will be blinded to study enrollment arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): The intervention consists of a brief contraception educational video and then the 10-week texting intervention which consists of 30 automated, personalized and interactive texting algorithms (3 texts per week).
  Interventions: Behavioral: Dr. Erica
- Control arm (No Intervention): Patients randomized to the control arm will receive the current standard discharge instructions provided in the investigator's ED.

INTERVENTIONS:
Behavioral: Dr. Erica — The 10 week texting intervention contains the follow characteristics to increase engagement: (1) Dr. ERICA (Emergency Room Interventions to Improve the Care of Adolescents): The persona and brand of the intervention is Dr. Erica, a relatable, empathetic, straightforward and reliable female doctor; (2) Personalization: Information collected at baseline will be incorporated into each individualized program; (3) Interactivity: The majority of text message algorithms contain 3-4 two-way automated messaging conversations. (4) Feedback loops: The investigators will collect feedback from participants to prompt action; (5) Visual stimuli: Texts include emojis, memes, and other visual stimuli, similar to current teen texting behaviors; (6) Social media: The investigators designed sexual health comic strips posted as an Instagram story; (7) Links and role modeling: Texts contain links to testimonials, influencers, and evidence-based websites.
  Arms: Intervention arm

SUMMARY:
This study will determine the feasibility, acceptability, and potential efficacy of an emergency department-based pregnancy prevention intervention targeting sexually active adolescent female emergency department patients.

DETAILED DESCRIPTION:
Emergency Departments (ED) care for 15 million adolescents each year. Adolescents who use the ED are at particularly high risk of unintended pregnancy. To date, no intervention has successfully increased contraception use among this high risk, hard-to-reach ED population.

In this study, the investigators will conduct a pilot randomized controlled trial of a user-informed, theory-based, personalized, interactive, pregnancy prevention text messaging intervention (Dr. Erica) to determine its feasibility, acceptability and potential efficacy. The investigators hypothesize that high risk adolescent female ED patients who receive Dr. Erica will more often initiate contraceptives than those females who receive standard discharge instructions alone.

At baseline and follow-up assessment at 3 months, participants will provide information regarding effective contraception initiation, any contraception at last intercourse, follow up with reproductive preventive health services, and contraception self-efficacy.

ELIGIBILITY:
Inclusion Criteria:

* female emergency department patient
* age 14-19 years
* sexually active with males in the past 3 months

Exclusion Criteria:

* currently using any effective form of contraception
* do not own a mobile phone with texting
* are pregnant
* are too ill for participation per the attending physician
* are cognitively impaired
* do not live locally
* do not speak English
* want to "become pregnant in the next year"

Ages: 14 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Female adolescent emergency department patients
Enrollment: 146 (Actual)
Dates: Start 2019-03-03 (Actual); Primary Completion 2020-07-02 (Actual); Study Completion 2020-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lauren S. Chernick, MD, MSc, Principal Investigator — Columbia University
Locations (1):
- Morgan Stanley Children's Hospital Emergency Department, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Arm | Control Arm
Started | 72 | 74
Completed | 59 | 64
Not Completed | 13 | 10

BASELINE CHARACTERISTICS:
Groups:
- Intervention Arm: Dr. Erica consists of two parts-a digital ED-based brief intervention and multimedia text messaging.
- Control Arm: Those randomized to usual care received an introductory text message to ensure texting capabilities for follow-up. No other edu- cation was provided outside usual care in the ED.
- Total: Total of all reporting groups
Arm/Group | Intervention Arm | Control Arm | Total
Number analyzed (Participants) | 72 | 74 | 146
Age, Customized [Count of Participants; unit: Participants]
  14-17 years old | 29 | 25 | 54
  18-19 years old | 43 | 49 | 92
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 74 | 146
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 20 | 14 | 34
  American Indian or Alaskan Native | 2 | 2 | 4
  White | 2 | 4 | 6
  Other | 39 | 40 | 79
  Unknown (data not collected) | 9 | 11 | 20
  Native American or Pacific Islander | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Potential Efficacy: Effective Contraception Initiation Rates [Time Frame: Enrollment, 12 Weeks Post-enrollment (2 Weeks Post Close of Intervention)]
Description: Initiation of effective contraception will be considered positive if participant self-reports initiation of effective contraception at follow up (telephone or online survey). An "effective" form of contraception (as defined by the World Health Organization) includes the following:
  * intrauterine device
  * birth control implant
  * birth control patch
  * birth control pills or oral contraceptives
  * injectable birth control
  * a vaginal ring
Time Frame: 3 months
Population: Only participants who provided self-report updates at the 3 months follow up mark were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 57 | 64
Participants | 14 | 14

2. Secondary Outcome: Feasibility: Percentage of Refusal
Description: Percentage of eligible participants who refused
Time Frame: Baseline
Population: Includes those who were eligible for enrollment who were screened for study participation.
Measure: Count of Participants; unit: Participants
Groups:
- All Those Eligible: All individuals who were considered to be eligible to participate in the study.
Arm/Group | All Those Eligible
Number analyzed (Participants) | 173
Participants | 27

3. Secondary Outcome: Feasibility: Opt Outs Measured Via Mobile Platform
Description: Percentage of enrolled participants in the intervention group who texted to stop receiving messages.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm
Number analyzed (Participants) | 72
Participants | 5

4. Secondary Outcome: Number of Enrolled Participants Who do Not Complete Follow up
Description: Measurement of the feasibility of Dr. Erica among adolescent female users
Time Frame: 3 months
Population: Includes the total number of participants randomized to each arm, regardless of follow up completion.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 72 | 74
Participants | 15 | 10

5. Secondary Outcome: Acceptability: Satisfaction With the Intervention Measured Via Online or Telephone Survey
Description: Percentage of participants in the intervention group who followed up and answered that they like the program and would recommend it to friends
Time Frame: 3 months
Population: Includes all participants in the intervention arm who completed the required follow up post-intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm
Number analyzed (Participants) | 49
Participants | 48

6. Secondary Outcome: Any Sex Over the Past 3 Months
Description: Self-report of any over the past 3 months.
Time Frame: 1 year
Population: Includes participants in each arm who completed the follow-up post-intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 49 | 59
Participants | 39 | 49

7. Other Pre Specified Outcome: Exploratory Efficacy Outcome: Number of Participants Who Followed up for Preventative Reproductive Care
Description: Participants who reported they did not go to the Columbia Family Planning Clinic over the past 3 months and answered "yes" to the question: "Over the past 3 months, have you seen a doctor for medical care?" In this Outcome, "preventative reproductive care" is defined as any visit to a doctor for the purposes of reproductive health.
Time Frame: 3 months
Population: This population answered "yes" or "no" the question prompted by Dr. Erica: "Over the past 3 months, have you been to the Columbia Family Planning Clinic?"
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 52 | 58
Participants | 35 | 42

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Intervention Arm | Control Arm
All-Cause Mortality (participants affected / at risk) | 0/72 | 0/74
Serious Adverse Events (participants affected / at risk) | 0/72 | 0/74
Other Adverse Events (participants affected / at risk) | 0/72 | 0/74

LIMITATIONS AND CAVEATS:
First, this study was conducted at a single center and represents a predominantly Hispanic population. Second, our intervention was available in only English. Third, participants did not respond to all follow-up questions, which may have affected our findings.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-01-08): https://cdn.clinicaltrials.gov/large-docs/11/NCT03866811/Prot_SAP_000.pdf
  • Informed Consent Form (2020-04-01): https://cdn.clinicaltrials.gov/large-docs/11/NCT03866811/ICF_001.pdf